CLINICAL TRIAL: NCT02202850
Title: Defining Which Remission Criterion At Month 6 Predicts Remission At Month 12 In A Real Life Clinical Practice, In A Cohort Of Ankylosing Spondylitis Patients Treated With Etanercept (Enbrel (Registered))
Brief Title: Defining Remission With Etanercept in AS in Real Life Clinical Practice
Acronym: REACH AS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801379; B1801379 (Other: Alias Study Number); REACH-AS (Other: Alias Study Number)
Record Dates: First submitted 2014-07-23; First posted 2014-07-29 (Estimated); Results first posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-04

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Etanercept First: Adults patients with AS receiving Etanercept as first biologic, according to prevailing reimbursement criteria in Belgium
  Interventions: Drug: etanercept
- Etanercept second: Adults patients with AS receiving Etanercept as second biologic, according to prevailing reimbursement criteria in Belgium
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — etanercept 1 x 50 mg/week or 2 x 25mg/week
  Groups: Etanercept First
Drug: etanercept — etanercept 1 x 50 mg/week or 2 x 25mg/week
  Groups: Etanercept second

SUMMARY:
Determine which remission criterion at Month 6 predicts remission at Month 12 the best.

DETAILED DESCRIPTION:
The analysis of the primary endpoint will be based on a logistic regression defining the dependent variable as the remission at Month 12 and the 6 independent variables as ASAS partial remission, ASAS 5/6, ASAS60, ASAS40, BASDAI50 and ASDAS inactive disease status.

This analysis will be conducted in each arm of the study as well as after a pooling of both patient groups.

In this context it seems reasonable to ensure the completion of the study by a total approximate number of 100 patients (approximately 50 patients per arm). In order to ensure 50 completers in each arm, 70 patients will be recruited at baseline, taking into account a drop-out rate of 30% over 1 year period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AS who start treatment with Etanercept according to prevailing reimbursement criteria and dosing in line with SmPC.

   1. First cohort: Etanercept is the first biological product prescribed
   2. Second cohort: Etanercept is the second biological product prescribed
2. Capable of understanding and willing to provide signed and dated written, voluntary informed consent before any protocol-specific procedures are performed.
3. 18 years of age or older at time of consent
4. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. History of or current psychiatric illness that would interfere with the subject's ability to comply with protocol requirements or to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting Rheumatologist for which the decision has been taken to prescribe Etanercept as first or second line
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2014-08-12 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- Belgium (29):
  - CHU Brugmann - Site Horta, Brussels, Bruxelles-capitale, Région de
  - ASZ Aalst, Aalst
  - Algemeen Stedelijk Ziekenhuis, Aalst
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Private Practice, Braine-l'Alleud
  - CHIREC, Brussels
  - CHU St-Pierre, Brussels
  - Private Practice, Champion
  - AZ Sint Blasius, Dendermonde
  - Private Practice, Flemalles Haute
  - Biomedical Research Institute/ Department of Rheumatology, Genk
  - Private Practice Rheumatology, Genk
  - ReumaClinic, Genk
  - Reumatologie Associatie, Genk
  - Private Practice, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - Grand Hopital de Charleroi, Gilly
  - Private Practice, Grand-Manil
  - AZ Groeninge Campus Sint Maarten, Kortrijk
  - CHU de Liège, Liège
  - Private Practice of Dr. Geert Ghyselen, Lokeren
  - Louisastraat 18, Mechelen
  - Hôpital Sainte Thérèse/ Department of Rheumatology, Montignies-sur-Sambre
  - Rheumatology, Ostend
  - Office of Maenaut Kristien, Schoten
  - Rheumatology, Sijsele-Damme
  - Sint-Andries Ziekenhuis, Tielt
  - Cliniques Universitaires UCL de Mont-Godinne, Yvoir

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801379&StudyName=Defining%20remission%20with%20etanercept%20in%20AS%20in%20real%20life%20clinical%20practice

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept First Cohort: Participants who had ankylosing spondylitis (AS) and commenced Etanercept as first biological product based on treating physician's discretion as per Summary of Product Characteristics (SmPC) and prevailing reimbursement criteria in Belgium, were observed prospectively for 12 months. According to SmPC, recommended dose included Etanercept 25 milligram (mg) twice weekly, 50 mg once weekly subcutaneous injection.
- Etanercept Second Cohort: Participants who had AS and commenced Etanercept as second biological product based on treating physician's discretion as per SmPC and prevailing reimbursement criteria in Belgium, were observed prospectively for 12 months. According to SmPC, recommended dose included Etanercept 25 mg twice weekly, 50 mg once weekly subcutaneous injection.
Period: Overall Study
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Started | 70 | 14
Completed | 46 | 8
Not Completed | 24 | 6
Not completed — Other | 2 | 2
Not completed — Enbrel treatment discontinued | 15 | 3
Not completed — Lost to Follow-up | 7 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis set (BAS) included all randomized participants enrolled in the study who were present at baseline, whether from first or second cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort | Total
Number analyzed (Participants) | 70 | 14 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.83 (13.84) | 41.37 (9.74) | 42.58 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 9 | 46
  Male | 33 | 5 | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Assessment of SpondyloArthritis International Society (ASAS) Partial Remission at Month 6 and Maintained Till Month 12
Description: ASAS partial remission was defined as a score of less than or equal to (<=) 2 for each of the 4 items including pain, function, participant global assessment (PGA) and inflammation. All these items were measured on a scale ranging from 0-10, where 0= no disease activity and 10= high disease activity.
Time Frame: Month 6 up to Month 12
Population: Completers analysis data set included all participants enrolled in the study, who completed the 12-month study, whether or not they missed some follow-up visits, and regardless of the cohort. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 34 | 5
percentage of participants | 14.7 [4.95 to 31.1] | 0.0 [0.0 to 52.2]

2. Primary Outcome: Percentage of Participants Who Achieved Assessment of SpondyloArthritis International Society (ASAS) 5/6 Remission Criteria at Month 6 and Maintained Till Month 12
Description: ASAS 5/6 was defined as at least greater than or equal to (>=) 20 percent relative improvement from baseline in at least 5 of the 6 following items: PGA, pain, function, inflammation, C - reactive protein (CRP) and spinal mobility. PGA, pain, function, inflammation all were measured on a scale ranging from 0-10, where 0= no disease activity and 10= high disease activity. CRP was measured in milligrams per liter (mg/L) and spinal mobility was measured in centimeter (cm) as calculated as the mean of right and left measurements of lateral spinal flexion.
Time Frame: Month 6 up to Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 30 | 5
percentage of participants | 43.3 [25.5 to 62.6] | 60.0 [14.7 to 94.7]

3. Primary Outcome: Percentage of Participants Who Achieved Assessment of SpondyloArthritis International Society (ASAS) 60 Remission Criteria at Month 6 and Maintained Till Month 12
Description: ASAS 60 was defined as at least >= 60 percent relative improvement from baseline and an absolute change >=2 scores in 3 of the 4 following items: PGA, pain, function, inflammation (where all were measured on a scale ranging from 0-10, where 0= no disease activity and 10= high disease activity) and no worsening in the remaining 2 domains: CRP (mg/L) and spinal mobility (cm).
Time Frame: Month 6 up to Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 34 | 5
percentage of participants | 29.4 [15.1 to 47.5] | 0.0 [0.0 to 52.2]

4. Primary Outcome: Percentage of Participants Who Achieved Assessment of SpondyloArthritis International Society (ASAS) 40 Remission Criteria at Month 6 and Maintained Till Month 12
Description: ASAS 40 was defined as at least >= 40 percent relative improvement from baseline and an absolute change >=2 scores in 3 of the 4 following items: PGA, pain, function, inflammation (where all were measured on a scale ranging from 0-10, where 0= no disease activity and 10= high disease activity) and no worsening in the remaining 2 domains: CRP (mg/L) and spinal mobility (cm).
Time Frame: Month 6 up to Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 34 | 5
percentage of participants | 32.4 [17.4 to 50.5] | 20.0 [0.51 to 71.6]

5. Primary Outcome: Percentage of Participants Who Achieved the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 Remission Criteria at Month 6 and Maintained Till Month 12
Description: BASDAI is a validated self-assessment tool used to determine disease activity in participant with AS by measuring participant's pain, discomfort and inflammation. Participant's pain, discomfort and inflammation was measured on a scale ranging from 0= none to 10= severe, where higher scores indicated higher degree of pain/discomfort/inflammation. The total BASDAI score was calculated as average of individual scores and ranged from 0= none to 10= severe, where higher score indicated high disease activity. BASDAI 50 remission was defined as at least >=50 percent relative improvement from baseline in BASDAI total score.
Time Frame: Month 6 up to Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 36 | 5
percentage of participants | 27.8 [14.2 to 45.2] | 0.0 [0.0 to 52.2]

6. Primary Outcome: Percentage of Participants Who Achieved the Ankylosing Spondylitis Disease Activity Score Based on C-Reactive Protein (ASDAS-CRP) Remission Criteria at Month 6 and Maintained Till Month 12
Description: ASDAS-CRP was based on 3 domains: BASDAI, Bath Ankylosing Spondylitis Global score (BAS-G) and CRP (in mg/L). BASDAI was used to measure disease activity by measuring participant's pain, discomfort and inflammation on a scale ranging from 0= none to 10= severe, where higher scores indicated higher degree of pain/discomfort/inflammation. The total BASDAI score was calculated as average of individual scores and ranged from 0= none to 10= severe, where higher score indicated lesser movement of participant due to AS. BAS-G was used to measure spinal pain on a scale ranging from 0= none to 10= severe, where higher scores indicated worsen health status. Scores from these 3 individual domains were averaged to calculate the ASDAS-CRP total scores. ASDAS-CRP remission was defined as having total ASDAS-CRP score of <1.3 on a scale ranging from 0= none to 10= severe, where higher scores indicated higher disease activity.
Time Frame: Month 6 up to Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 28 | 5
percentage of participants | 10.7 [2.27 to 28.2] | 0.0 [0.0 to 52.2]

7. Primary Outcome: Percentage of Participants Who Achieved the Ankylosing Spondylitis Disease Activity Score Based on Erythrocyte Sedimentation Rate (ASDAS-ESR) Remission Criteria at Month 6 and Maintained Till Month 12
Description: ASDAS-ESR was based on 3 domains: BASDAI, BAS-G and ESR (in millimeter per hour). BASDAI was used to measure disease activity by measuring participant's pain, discomfort and inflammation on a scale ranging from 0= none to 10= severe, where higher scores indicated higher degree of pain/discomfort/inflammation. The total BASDAI score was calculated as average of individual scores and ranged from 0= none to 10= severe, where higher score indicated lesser movement of participant due to AS. BAS-G was used to measure spinal pain on a scale ranging from 0= none to 10= severe, where higher scores indicated worsen health status. Scores from these 3 individual domains were averaged to calculate the ASDAS- ESR total scores. ASDAS- ESR remission was defined as having total ASDAS- ESR score of <1.3 on a scale ranging from 0= none to 10= severe, where higher scores indicated higher disease activity.
Time Frame: Month 6 up to Month 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 20 | 4
percentage of participants | 15.0 [3.21 to 37.9] | 0.0 [0.0 to 52.2]

8. Secondary Outcome: Percentage of Participants Who Achieved Assessment of SpondyloArthritis International Society (ASAS) Partial Remission Criteria at Month 3, 6, 9 and 12
Description: ASAS partial remission was defined as a score of <= 2 for each of the 4 items including pain, function, PGA and inflammation. All these items were measured on a scale ranging from 0-10, where 0= no disease activity and 10= high disease activity.
Time Frame: Month 3, 6, 9 and 12
Population: Completers analysis data set included all participants enrolled in the study, who completed the 12-month study, whether or not they missed some follow-up visits, and regardless of the cohort.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 46 | 8
percentage of participants
  Month 3: number analyzed (Participants) | 40 | 7
  Month 3 | 12.5 [4.19 to 26.8] | 0.0 [0.0 to 41.0]
  Month 6: number analyzed (Participants) | 34 | 5
  Month 6 | 17.7 [6.76 to 34.5] | 0.0 [0.0 to 52.2]
  Month 9: number analyzed (Participants) | 30 | 6
  Month 9 | 16.7 [5.64 to 34.7] | 0.0 [0.0 to 45.9]
  Month 12: number analyzed (Participants) | 42 | 7
  Month 12 | 21.4 [10.3 to 36.8] | 14.3 [0.36 to 57.9]

9. Secondary Outcome: Percentage of Participants Who Achieved Assessment of SpondyloArthritis International Society (ASAS) 5/6 Remission Criteria at Month 3, 6, 9 and 12
Description: ASAS 5/6 was defined as at least >= 20 percent relative improvement from baseline in at least 5 of the 6 following items: PGA, pain, function, inflammation, CRP and spinal mobility. PGA, pain, function, inflammation all were measured on a scale ranging from 0-10, where 0= no disease activity and 10= high disease activity. CRP was measured in mg/L and spinal mobility was measured in centimeter as calculated as the mean of right and left measurements of lateral spinal flexion.
Time Frame: Month 3, 6, 9 and 12
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 46 | 8
percentage of participants
  Month 3: number analyzed (Participants) | 35 | 5
  Month 3 | 51.4 [34.0 to 68.6] | 20.0 [0.51 to 71.6]
  Month 6: number analyzed (Participants) | 30 | 5
  Month 6 | 46.7 [28.3 to 65.7] | 60.0 [14.7 to 94.7]
  Month 9: number analyzed (Participants) | 26 | 6
  Month 9 | 57.7 [36.9 to 76.7] | 33.3 [4.33 to 77.7]
  Month 12: number analyzed (Participants) | 39 | 5
  Month 12 | 61.5 [44.6 to 76.6] | 60.0 [14.7 to 97.7]

10. Secondary Outcome: Percentage of Participants Who Achieved Assessment of SpondyloArthritis International Society (ASAS) 60 Remission Criteria at Month 3, 6, 9 and 12
Description: as for outcome 3
Time Frame: Month 3, 6, 9 and 12
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 46 | 8
percentage of participants
  Month 3: number analyzed (Participants) | 40 | 7
  Month 3 | 30.0 [16.6 to 46.5] | 0.0 [0.0 to 41.0]
  Month 6: number analyzed (Participants) | 34 | 5
  Month 6 | 32.4 [17.4 to 50.5] | 0.0 [0.0 to 52.2]
  Month 9: number analyzed (Participants) | 30 | 6
  Month 9 | 33.3 [17.3 to 52.8] | 0.0 [0.0 to 45.9]
  Month 12: number analyzed (Participants) | 41 | 7
  Month 12 | 29.3 [16.1 to 45.5] | 14.3 [0.36 to 57.9]

11. Secondary Outcome: Percentage of Participants Who Achieved Assessment of SpondyloArthritis International Society (ASAS) 40 Remission Criteria at Month 3, 6, 9 and 12
Description: as for outcome 4
Time Frame: Month 3, 6, 9 and 12
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 46 | 8
percentage of participants
  Month 3: number analyzed (Participants) | 40 | 7
  Month 3 | 37.5 [22.7 to 54.2] | 28.6 [3.67 to 71.0]
  Month 6: number analyzed (Participants) | 34 | 5
  Month 6 | 41.2 [24.7 to 59.3] | 20.0 [0.51 to 71.6]
  Month 9: number analyzed (Participants) | 30 | 6
  Month 9 | 46.7 [28.3 to 65.7] | 16.7 [0.42 to 64.1]
  Month 12: number analyzed (Participants) | 41 | 7
  Month 12 | 46.3 [30.7 to 62.6] | 42.9 [9.90 to 81.6]

12. Secondary Outcome: Percentage of Participants Who Achieved the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 Remission Criteria at Month 3, 6, 9 and 12
Description: as for outcome 5
Time Frame: Month 3, 6, 9 and 12
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 46 | 8
percentage of participants
  Month 3: number analyzed (Participants) | 41 | 7
  Month 3 | 41.5 [26.3 to 57.9] | 14.3 [0.36 to 57.9]
  Month 6: number analyzed (Participants) | 36 | 5
  Month 6 | 30.6 [16.4 to 48.1] | 0.0 [0.00 to 52.2]
  Month 9: number analyzed (Participants) | 31 | 6
  Month 9 | 45.2 [27.3 to 64.0] | 0.0 [0.0 to 45.9]
  Month 12: number analyzed (Participants) | 45 | 8
  Month 12 | 42.2 [27.7 to 57.9] | 25.0 [3.19 to 65.1]

13. Secondary Outcome: Percentage of Participants Who Achieved the Ankylosing Spondylitis Disease Activity Score Based on C-Reactive Protein (ASDAS-CRP) Remission Criteria at Month 3, 6, 9 and 12
Description: ASDAS-CRP was based on 3 domains: BASDAI, BAS-G and CRP (in mg/L). BASDAI was used to measure disease activity by measuring participant's pain, discomfort and inflammation on a scale ranging from 0= none to 10= severe, where higher scores indicated higher degree of pain/discomfort/inflammation. The total BASDAI score was calculated as average of individual scores and ranged from 0= none to 10= severe, where higher score indicated lesser movement of participant due to AS. BAS-G was used to measure spinal pain on a scale ranging from 0= none to 10= severe, where higher scores indicated worsen health status. Scores from these 3 individual domains were averaged to calculate the ASDAS-CRP total scores. ASDAS-CRP remission was defined as having total ASDAS-CRP score of <1.3 on a scale ranging from 0= none to 10= severe, where higher scores indicated higher disease activity.
Time Frame: Month 3, 6, 9 and 12
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 46 | 8
percentage of participants
  Month 3: number analyzed (Participants) | 33 | 5
  Month 3 | 24.2 [11.1 to 42.3] | 0.0 [0.0 to 52.2]
  Month 6: number analyzed (Participants) | 28 | 5
  Month 6 | 17.9 [6.06 to 36.9] | 0.0 [0.0 to 52.2]
  Month 9: number analyzed (Participants) | 23 | 5
  Month 9 | 26.1 [10.2 to 48.4] | 0.0 [0.0 to 52.2]
  Month 12: number analyzed (Participants) | 39 | 6
  Month 12 | 30.8 [17.0 to 47.6] | 0.0 [0.0 to 45.9]

14. Secondary Outcome: Percentage of Participants Who Achieved the Ankylosing Spondylitis Disease Activity Score Based on Erythrocyte Sedimentation Rate (ASDAS-ESR) Remission Criteria at Month 3, 6, 9 and 12
Description: as for outcome 7
Time Frame: Month 3, 6, 9 and 12
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 46 | 8
percentage of participants
  Month 3: number analyzed (Participants) | 25 | 5
  Month 3 | 16.0 [4.54 to 36.1] | 0.0 [0.0 to 52.2]
  Month 6: number analyzed (Participants) | 20 | 4
  Month 6 | 20.0 [5.73 to 43.7] | 0.0 [0.0 to 60.2]
  Month 9: number analyzed (Participants) | 13 | 4
  Month 9 | 15.4 [1.92 to 45.5] | 0.0 [0.0 to 60.2]
  Month 12: number analyzed (Participants) | 31 | 5
  Month 12 | 19.4 [7.45 to 37.5] | 20.0 [0.51 to 71.6]

15. Secondary Outcome: Change From Baseline in Participant Global Assessment (PGA) Score at Month 6 and 12
Description: Participants were asked to assess their disease activity on an 11-point scale of 0 (no disease activity) to 10 (extreme disease activity), where higher score indicated higher disease activity.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 46 | 8
Units on a scale
  Baseline | 7.61 (1.78) | 7.63 (0.92)
  Change at Month 6: number analyzed (Participants) | 34 | 5
  Change at Month 6 | 3.62 (2.81) | 2.60 (2.30)
  Change at Month 12: number analyzed (Participants) | 42 | 7
  Change at Month 12 | 3.43 (2.96) | 3.00 (2.00)

16. Secondary Outcome: Change From Baseline in Pain Score of Ankylosing Spondylitis at Month 6 and 12
Description: Pain score is used to determine disease activity in participants with AS by measuring participants pain and swelling, on a scale ranging from 0= none to 10= severe, where higher scores indicated higher degree of pain/swelling. The total pain score was calculated as average of these 2 items and ranged from 0= none to 10= severe, where higher score indicated higher degree of pain in participant due to AS.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 46 | 8
Units on a scale
  Baseline | 6.40 (2.05) | 7.00 (1.39)
  Change at Month 6: number analyzed (Participants) | 36 | 5
  Change at Month 6 | 2.15 (2.61) | 1.70 (1.57)
  Change at Month 12: number analyzed (Participants) | 45 | 8
  Change at Month 12 | 2.60 (2.96) | 2.81 (2.17)

17. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) Score at Month 6 and 12
Description: BASFI was a functional index which included 10 items assessing ability of participants to perform normal daily activities. Each item was scored on a scale of 0=easy, to 10=impossible. The BASFI total score was calculated as the average score of these 10 individual items. BASFI total score ranged from 0 to 10, where higher scores indicated more severe disease activity.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 46 | 8
Units on a scale
  Baseline | 5.90 (2.35) | 7.34 (1.15)
  Change at Month 6: number analyzed (Participants) | 36 | 5
  Change at Month 6 | 2.07 (2.50) | 1.90 (0.47)
  Change at Month 12: number analyzed (Participants) | 44 | 8
  Change at Month 12 | 2.15 (2.65) | 2.39 (2.28)

18. Secondary Outcome: Change From Baseline in Inflammation Score of Ankylosing Spondylitis at Month 6 and 12
Description: Inflammation score is used to determine disease activity in participants with AS by measuring intensity and duration of inflammation, on a scale ranging from 0= none to 10= severe, where higher scores indicated higher degree of inflammation. The total inflammation score was calculated as average of these 2 items and ranged from 0= none to 10= severe, where higher score indicated higher degree of inflammation in participant due to AS.
Time Frame: Baseline, Month 6 and12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 46 | 8
Units on a scale
  Baseline | 5.98 (2.24) | 6.81 (1.56)
  Change at Month 6: number analyzed (Participants) | 36 | 5
  Change at Month 6 | 2.71 (2.34) | 3.40 (1.95)
  Change at Month 12: number analyzed (Participants) | 45 | 8
  Change at Month 12 | 3.07 (2.60) | 2.50 (2.19)

19. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) at Month 6 and 12
Description: CRP is a protein marker in the blood for inflammation.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milligrams per liter
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 46 | 8
milligrams per liter
  Baseline: number analyzed (Participants) | 45 | 8
  Baseline | 14.49 (14.14) | 6.06 (4.83)
  Change at Month 6: number analyzed (Participants) | 30 | 5
  Change at Month 6 | 1.45 (46.86) | 5.04 (1.28)
  Change at Month 12: number analyzed (Participants) | 41 | 6
  Change at Month 12 | 11.50 (14.70) | -2.03 (9.47)

20. Secondary Outcome: Change From Baseline in Spinal Mobility Measurement at Month 6 and 12
Description: Spinal mobility was the mean of right and left measurements of lateral spinal flexion in centimeters.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 46 | 8
centimeters
  Baseline: number analyzed (Participants) | 35 | 6
  Baseline | 10.04 (4.87) | 10.80 (4.51)
  Change at Month 6: number analyzed (Participants) | 18 | 3
  Change at Month 6 | -3.13 (3.41) | -0.83 (3.82)
  Change at Month 12: number analyzed (Participants) | 27 | 4
  Change at Month 12 | -3.73 (5.30) | 1.08 (4.68)

21. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Month 6 and 12
Description: BASDAI is a validated self-assessment tool used to determine disease activity in participant with AS by measuring participant's pain, discomfort and inflammation. Participant's pain, discomfort and inflammation was measured on a scale ranging from 0= none to 10= severe, where higher scores indicated higher degree of pain/discomfort/inflammation. The total BASDAI score was calculated as average of individual scores and ranged from 0= none to 10= severe, where higher score indicated high disease activity.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 46 | 8
Units on a scale
  Baseline | 6.45 (1.61) | 7.14 (0.90)
  Change at Month 6: number analyzed (Participants) | 36 | 5
  Change at Month 6 | 2.16 (2.36) | 2.16 (1.47)
  Change at Month 12: number analyzed (Participants) | 45 | 8
  Change at Month 12 | 2.62 (2.53) | 2.48 (2.05)

22. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score Based on C-Reactive Protein (ASDAS-CRP) at Month 6 and 12
Description: as for outcome 13
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 46 | 8
Units on a scale
  Baseline: number analyzed (Participants) | 45 | 8
  Baseline | 3.73 (0.86) | 3.54 (0.87)
  Change at Month 6: number analyzed (Participants) | 28 | 5
  Change at Month 6 | 1.44 (1.06) | 1.54 (0.61)
  Change at Month 12: number analyzed (Participants) | 39 | 6
  Change at Month 12 | 1.70 (1.15) | 1.17 (1.01)

23. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score Based on Erythrocyte Sedimentation Rate (ASDAS-ESR) at Month 6 and 12
Description: as for outcome 7
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
Number analyzed (Participants) | 46 | 8
Units on a scale
  Baseline: number analyzed (Participants) | 33 | 7
  Baseline | 3.25 (0.75) | 3.51 (0.69)
  Change at Month 6: number analyzed (Participants) | 16 | 4
  Change at Month 6 | 1.17 (0.65) | 1.11 (0.45)
  Change at Month 12: number analyzed (Participants) | 26 | 5
  Change at Month 12 | 1.18 (0.87) | 1.25 (0.94)

ADVERSE EVENTS:
Time Frame: Baseline up to Month 12
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Etanercept First Cohort | Etanercept Second Cohort
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/14
Serious Adverse Events (participants affected / at risk) | 3/70 | 0/14
Other Adverse Events (participants affected / at risk) | 18/70 | 2/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept First Cohort (N=70) | Etanercept Second Cohort (N=14)
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Etanercept First Cohort (N=70) | Etanercept Second Cohort (N=14)
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Injection site hypersensitivity (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Injection site inflammation (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Injection Site Erythema (General disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paresthesia (Nervous system disorders) | 2 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1/37 | 0/9 — This event was gender specific.
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Large Intestinal Polypectomy (Surgical and medical procedures) | 1 | 0
Uveitis (Eye disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT02202850/Prot_SAP_000.pdf